CLINICAL TRIAL: NCT07332949
Title: Impact of Dialysis on Sexuality.
Acronym: SEXODIA
Status: Recruiting | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/04; 2025-A02271-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2025-12-19; First posted 2026-01-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Hemodialysis; Peritoneal dialysis; Sexuality
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults treated with chronic dialysis
  Interventions: Other: Questionnaire on sexuality

INTERVENTIONS:
Other: Questionnaire on sexuality — The patients will receive the following questionnaires to complete during the dialysis session:
  * MSHQ (Male Sexual Health Questionnaire) for men
  * FSFI (Female Sexual Function Index) for women Additional questions addressing medical history and body image perception are included.

SUMMARY:
Sexuality is an essential dimension of quality of life and is frequently impaired in patients with end-stage chronic kidney disease undergoing hemodialysis. Sexual dysfunctions-including erectile dysfunction, reduced sexual desire, and difficulties with arousal or orgasm-are highly prevalent in this population. These disorders have multifactorial origins, involving hormonal disturbances, comorbidities, treatment-related side effects, chronic fatigue, and the psychological and relational impact of long-term illness.

Despite their frequency, sexual health issues are rarely addressed in routine dialysis care. This is largely due to time constraints during consultations, insufficient training of healthcare professionals, and persistent social and cultural taboos. In addition, the existing scientific literature remains limited, often outdated, and predominantly focused on male patients. Data concerning women, sexual diversity, body image, and couple-related aspects are scarce. Standard kidney disease-specific quality-of-life instruments, such as the KDQOL questionnaire, provide only a minimal assessment of sexuality, with a single item related to sexual desire.

The aim of this study is to provide a contemporary and comprehensive assessment of the impact of dialysis on sexual quality of life. By documenting sexual function and sexual complaints in patients undergoing dialysis, this study seeks to improve understanding of patients' experiences and to facilitate communication between patients and healthcare professionals. Ultimately, the findings are intended to support better integration of sexual health into routine nephrology care and to contribute to improved clinical practices in the field of sexual health.

This study is designed as a cross-sectional survey conducted among patients undergoing dialysis at the Groupe Hospitalier Privé Ambroise Paré-Hartmann in the Paris area. Eligible patients are informed about the study during a dialysis session by a healthcare professional (dialysis nurse, nephrologist, or physiotherapist specialized in sexology). Participants complete a self-administered questionnaire during their dialysis session, including the Male Sexual Health Questionnaire (MSHQ) for men and the Female Sexual Function Index (FSFI) for women. Additional questions addressing medical history and body image perception are included. The estimated completion time for the questionnaire is approximately 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years,
* Treated with chronic dialysis (hemodialysis or peritoneal dialysis) for at least 6 months.

Exclusion Criteria:

* Major cognitive or psychiatric disorders that make understanding or completing the questionnaire difficult.
* General health condition not allowing participation without significant discomfort or excessive fatigue.
* Opposition by the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults treated with chronic dialysis (hemodialysis or peritoneal dialysis).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Sexual quality of life | At baseline, during a dialysis session
  The MSHQ questionnaire for men consists of 25 questions, minimum score: 25, maximum score: 125. A higher score on this scale indicates better sexual function.
Sexual quality of life | At baseline, during a dialysis session
  The FSFI questionnaire for women consists of 19 questions, minimum score: 2, maximum score: 36. A higher score on this scale indicates better sexual function.

SECONDARY OUTCOMES:
Body perception | At baseline, during a dialysis session
  Questionnaire adapted from the Body Image Scale consisting of 4 questions, minimum score: 0, maximum score: 12. A higher score indicates a poorer body image.

CONTACTS AND LOCATIONS:
Locations (1):
- Ambroise Paré - Hartmann Private Hospital Group, Neuilly-sur-Seine, Île-de-France Region, France